CLINICAL TRIAL: NCT06978192
Title: The Clinical Efficacy Analysis of Long-Duration High-Voltage Pulsed Radiofrequency Combined With Dexmedetomidine Nasal Spray in the Treatment of Herpes Zoster-Associated Neuropathic Pain
Brief Title: Clinical Study on the Treatment of Herpes Zoster Pain With Dexmedetomidine Combined With Long-term High Voltage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fenghui Deng (Other)
Responsible Party: Sponsor-Investigator, Fenghui Deng, Associate chief of pain, Zunyi Medical College
Organization: Zunyi Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KLLY-2024-235
Record Dates: First submitted 2025-04-16; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Herpes Zoster (HZ)
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HL-PRF +DNS (Experimental): On the basis of conventional drug treatment, dexmedetomidine nasal spray was administered before HL-PRF treatment, before bedtime on the day of the operation, and before bedtime on the 1st to 3rd days after the operation.
  Interventions: Drug: dexmedetomidine nasal spray group; Other: long duration high voltage pulse RF therapy group
- HL-PRF (Other): on the basis of conventional drug treatment, and the long-duration high-voltage pulse radiofrequency therapy was performed.
  Interventions: Other: long duration high voltage pulse RF therapy group

INTERVENTIONS:
Drug: dexmedetomidine nasal spray group — Experimental group: Long duration high voltage pulse RF therapy plus dexmedetomidine nasal spray group
  Arms: HL-PRF +DNS
Other: long duration high voltage pulse RF therapy group — Experimental group: long duration high voltage pulse RF therapy group

SUMMARY:
Participants will be invited to take part in clinical research. This informed consent form will provide information to the participants to help them decide whether to participate in the clinical study. If participants have any questions, please ask them directly to the researcher in charge of this study. This study was approved by the Biomedical Research Ethics Review Committee of the Institute. This trial is a randomized controlled clinical study. According to the different treatment methods, the control group was randomly divided into the control group and the experimental group. Control group: On the basis of conventional drug treatment, long-term high-voltage pulsed radiofrequency treatment was carried out. Experimental group: On the basis of conventional drug treatment, dexmedetomidine nasal spray was administered before HL-PRF treatment, before bedtime on the day of the operation, and before bedtime on the 1st to 3rd days after the operation. Heart rate, blood pressure and blood oxygen saturation were monitored respectively before the operation, during the operation and after the operation. Telephone follow-ups were conducted at 1 week, 1 month, 3 months and 6 months after the operation respectively. If the participants agree to participate in this study, the researchers will number the participants and establish medical records. The researchers will have detailed communication with the participants or their families, inform them of the research situation, and ask the participants to provide disease information, including the onset of the disease, family history, previous medical visits and some examination results.

What do you need to do in this research? Once participating in the study, participants will be required to provide true information about their medical history and current physical condition. Tell the research doctor about any discomfort you encountered during the research process; Do not take restricted drugs, foods, etc. Tell the research doctor whether you have participated in or are currently participating in any other research recently.

Risks and discomfort: Communicating and talking with researchers may cause participants to feel psychologically uncomfortable.

Since this study only collected the medical history, data and epidemiological investigation of patients or normal people, there is no harm in this study. If participants are injured during the clinical trial, they can receive free treatment and/or appropriate compensation in accordance with Chinese law.

What are the benefits of participating in this research? Useful information can be provided for disease research by studying the information of the participants.

The cost of participating in this study: Participation in this study will be based on the medical information of the research participants, and the related costs will not be borne by the participants.

Privacy issue: If participants decide to take part in this study, their participation status and personal data during the study period will be kept confidential. When necessary, government administrative departments or members of the ethics review committee may access the personal data of participants in research institutions. When the results of this study are announced, the personal identity information of the participants will not be disclosed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adverse reactions that are not effective in conventional drug treatment and cannot tolerate drugs
* The pain is located in the corresponding innervated are
* The pain affects the patient's daily life or work
* Diagnostic nerve block is effective and pain limited
* Recurrent herpes zoster pain
* Patients with shingle-related pain aged 40-85 years

Exclusion Criteria:

* Infection at the puncture site, systemic infection that may spread, and malignant tumors near the puncture
* There are contraindications in minimally invasive interventional therapy such as coagulation function and platelet dysfunction
* Allergies to local anesthetics and inhalants
* Heart, lung, liver, kidney and other important organ failure, can not tolerate surgery
* Severe endocrine system diseases or long-term use of hormone or immunosuppressive therapy
* Patients with cardiac pacemakers, pregnant or lactating women
* Patients with cognitive dysfunction or poor coordination
* Patients who have been treated with electrical stimulation or PRF

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NRS) | The patients were evaluated respectively before the operation, on the 7th day, the 30th day, the 90th day and the 180th day after the operation.
  The pain degree of the patients was evaluated by using the Numerical Rating Scale for Pain (NRS). The NRS score was 0 when there was no pain. 1 to 3 points indicate mild pain. Points 4 to 6 indicate moderate pain. A score of 7 to 10 indicates severe pain.
The Hamilton Anxiety Scale (HAMA) | The scores were evaluated respectively before the operation, 7 days after the operation, 30 days after the operation, 90 days after the operation and 180 days after the operation.
  uses a 5-point scoring system ranging from 0 to 4. A total score of ≥29 points may indicate severe anxiety. A score of 21 or above definitely indicates obvious anxiety. A score of 14 or above definitely indicates anxiety. A score above 7 May indicate anxiety. If it is less than 7 points, there will be no anxiety symptoms.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | The PSQI scores were recorded respectively before the operation, on the 7th day, 30th day, 90th day and 180th day after the operation.
  The total PSQI score is between 0 and 20 points. The lower the score is, the better the sleep quality will be
Interleukin 6 | Before the operation and the first day after the operation.
  Interleukin-6 (IL-6) levels are positively correlated with the severity of postherpetic neuralgia (PHN) pain.
blood pressure | Before, during and immediately after the operation
  Measure blood pressure and record systolic and diastolic blood pressure respectively, with the unit being mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Deng, Principal Investigator — Fenghui
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No